CLINICAL TRIAL: NCT01765426
Title: Phase 1b, Partial-Blind, Parallel Group, Randomized Study to Investigate the Safety and Immunogenicity of a Tetravalent Chimeric Dengue Vaccine (DENVax) Administered Intradermally Using Needle or a Needle-Free PharmaJet® Injector in Healthy Adults
Brief Title: Phase 1b Study Investigating Safety & Immunogenicity of TDV Given Intradermally by Needle or Needle-Free PharmaJet Injector
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11-0049; U1111-1178-6503 (Registry Identifier: WHO)
Record Dates: First submitted 2012-12-17; First posted 2013-01-10 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers
Keywords: Prophylactic vaccination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: TDV using PharmaJet® Injector (Experimental): Takeda's Tetravalent Dengue Vaccine Candidate (TDV) [previously DENVax] one dose injection in arm 1 and placebo: phosphate buffered saline (PBS) one dose injection in arm 2, using needle-free PharmaJet® Injector, intradermal, on Day 0 and TDV, injection using needle-free PharmaJet® Injector, intradermal, one dose on Day 90.
  Interventions: Biological: TDV; Drug: Placebo
- Group 2: TDV using PharmaJet® Injector (Experimental): TDV injection, one dose in each arm, using needle-free PharmaJet® Injector, intradermal, on Day 0 and placebo: PBS, injection using needle-free PharmaJet® Injector, intradermal, one dose on Day 90.
  Interventions: Biological: TDV; Drug: Placebo
- Group 3: TDV using Needle and Syringe (Experimental): TDV one dose injection in arm 1 and placebo: PBS one dose injection in arm 2, using needle and syringe, intradermal, on Day 0 and TDV injection using needle and syringe, intradermal, one dose on Day 90.
  Interventions: Biological: TDV; Drug: Placebo
- Group 4: TDV using PharmaJet® Injector (Experimental): TDV injection, one dose in each arm, using needle-free PharmaJet® Injector, intradermal, on Day 0 and TDV, injection using needle-free PharmaJet® Injector, intradermal, one dose on Day 90.
  Interventions: Biological: TDV

INTERVENTIONS:
Biological: TDV — TDV suspension for intradermal administration
Drug: Placebo — Phosphate buffered saline (PBS)
  Arms: Group 1: TDV using PharmaJet® Injector; Group 2: TDV using PharmaJet® Injector; Group 3: TDV using Needle and Syringe

SUMMARY:
The purpose of this study is to compare the safety, tolerability and immunogenicity of Takeda's Tetravalent Dengue Vaccine Candidate (TDV) [previously DENVax] when administered intradermally in varied dosing schedules and via different methods of administration (conventional needle/syringe versus needle-free PharmaJet® injector).

DETAILED DESCRIPTION:
This is an exploratory trial to assess the safety, tolerability and immunogenicity of vaccination with a tetravalent dengue vaccine (TDV) in healthy adults delivered intradermally using the conventional needle/syringe or a needle-free PharmaJet® injector.

Two (2) intradermal injections of either vaccine or placebo will be administered to qualified participants (one in each arm) on Day 0 of the study. A subsequent injection will also be given on Day 90 with either vaccine or placebo (in one arm only).

Participants will be evaluated for safety and dengue neutralizing antibody to all four serotypes. All participants will also be evaluated for injection site reactions and have blood drawn for viremia, neutralizing antibodies, cell mediated immunity and innate immunity.

Participants will be required to participate for approximately 10 months from recruitment and collection of data for primary outcomes (through Day 120) including collection of additional samples for measurement of longer term antibody titers (through Day 270).

This project has been funded in whole or in part with Federal funds from the National Institute of Allergy and Infectious Diseases, National Institutes of Health, Department of Health and Human Services, under Contract No. HHSN272201000034C.

ELIGIBILITY:
Inclusion Criteria:

* In good health as determined by medical history and physical examination (including blood pressure and heart rate).
* Negative for human immunodeficiency virus-1 (HIV-1) antibodies, Hepatitis C antibodies & Hepatitis B surface antigen.
* Females negative by urine pregnancy test at screening and immediately prior to injection, and were willing to use reliable means of contraception.
* Body Mass Index (BMI) ≤ 35 kg/m^2.

Exclusion Criteria:

* Any Grade 2 or above abnormality in the screening laboratory tests.
* History of Dengue Fever, Japanese Encephalitis, West Nile or Yellow Fever disease.
* Seropositivity to dengue or West Nile virus.
* Extensive scarring or tattoo (> 50%) on arms, shoulders, neck face and head.
* History of significant dermatologic disease in the last 6 months.
* Receipt or planned receipt of any vaccine in the 4 weeks preceding or following the Day 0 or 90 vaccinations.
* Any planned travel to dengue endemic areas including the Caribbean, Mexico, Central America, South America or Southeast Asia, during the study period and during the month prior to screening.
* Use of systemic corticosteroids therapy within the previous 6 months (at a dose of 0.5 mg/kg/day). Topical prednisone is not permitted if currently in use or used within the last month prior to the first vaccination.
* Use of any prescribed medication 7 days before the first injection.
* Previous vaccination in a clinical study or with an approved product against Dengue Fever, Yellow Fever and or Japanese Encephalitis.
* Known or suspected congenital or acquired immunodeficiency or receipt of immunosuppressive therapy in the last 6 months.
* Planned donation of blood during the period of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2013-02-15 (Actual); Primary Completion 2014-06-26 (Actual); Study Completion 2014-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (2):
- United States (2):
  - University of Texas Medical Branch, Galveston, Texas
  - Group Health Research Institute, Seattle, Washington

REFERENCES:
- [Derived] Jackson LA, Rupp R, Papadimitriou A, Wallace D, Raanan M, Moss KJ. A phase 1 study of safety and immunogenicity following intradermal administration of a tetravalent dengue vaccine candidate. Vaccine. 2018 Jun 22;36(27):3976-3983. doi: 10.1016/j.vaccine.2018.05.028. Epub 2018 May 19. PMID 29789238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 15 February 2013 (First participant signed Informed Consent Form) to 26 June 2014 (date of last participant's visit/contact).
Pre-assignment Details: Healthy Volunteers were enrolled equally in 1 of 4 treatment groups: Group 1 (2 doses), Group 2 (2 doses) Group 4 (3 doses) of Tetravalent Dengue Vaccine (TDV) using PharmaJet® Injector and Group 3 (2 doses) TDV using needle and syringe.
Period: Overall Study
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Started | 18 | 17 | 17 | 15
Completed All Vaccinations | 17 | 16 | 17 | 15
Completed | 18 | 16 | 17 | 15
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector | Total
Number analyzed (Participants) | 18 | 17 | 17 | 15 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (8.47) | 32.4 (8.87) | 30.1 (7.90) | 27.5 (6.84) | 29.9 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 5 | 9 | 26
  Male | 13 | 10 | 12 | 6 | 41
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 1 | 0 | 0 | 3 | 4
  Non-Hispanic | 17 | 17 | 17 | 12 | 63
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 1 | 2 | 0 | 4
  Black or African American | 4 | 0 | 0 | 1 | 5
  White | 13 | 14 | 13 | 12 | 52
  Multi-Racial | 0 | 1 | 2 | 2 | 5
  Other | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 17 | 15 | 67
Weight [Mean (Standard Deviation); unit: kg] | 78.77 (20.349) | 81.19 (15.673) | 76.72 (13.672) | 73.73 (8.939) | 77.73 (15.354)
Height [Mean (Standard Deviation); unit: cm] | 174.47 (8.934) | 177.58 (9.891) | 179.77 (8.833) | 169.13 (10.593) | 175.41 (10.114)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.89 (6.458) | 25.73 (4.516) | 23.66 (3.406) | 25.93 (3.743) | 25.29 (4.733)
Seropositivity Status at Baseline [Number; unit: participants]
  Seropositive | 1 | 4 | 1 | 2 | 8
  Seronegative | 17 | 13 | 16 | 13 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local (Injection Site) Adverse Events (AEs) After Either Vaccine Dose by Maximum Severity as Assessed by the Clinical Staff
Description: An AE is defined as any untoward medical occurrence in a patient or clinical trial participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Local injection site reactions were evaluated by the blinded clinical staff and include: erythema (redness), edema/induration (swelling), pain and pruritus (itching). Severity grades for erythema and edema are derived based on the Division of Microbiology and Infectious Diseases (DMID) toxicity grading longest diameters using the scale 0=none, 1=<15 millimeters (mm), 2=15 to 30 mm and 3=>30 mm (severe). Pain and itching were graded using the scale: 0=none to 4=requires ER visit or hospitalization. Local injection site reactions are presented as the percentage of participants experiencing a reaction, by reaction type, overall and by severity, using the participant's worst reported severity grade. Only categories for which there was at least 1 participant are reported.
Time Frame: 28 Days after each dose
Population: Safety analysis set included all randomized participants who received at least 1 dose of study vaccine (or placebo), including a partial dose.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Number analyzed (Participants) | 18 | 17 | 17 | 15
percentage of participants
  Edema, Grade 0 (None) | 16.7 | 11.8 | 11.8 | 13.3
  Edema, Any Severity >Grade 0 | 83.3 | 88.2 | 88.2 | 86.7
  Edema, Grade 1 (Mild) | 77.8 | 82.4 | 76.5 | 66.7
  Edema, Grade 2 (Moderate) | 5.6 | 5.9 | 11.8 | 20.0
  Erythema, Grade 0 (None) | 11.1 | 0 | 0 | 6.7
  Erythema, Any Severity >Grade 0 | 88.9 | 100.0 | 100.0 | 93.3
  Erythema, Grade 1 (Mild) | 55.6 | 23.5 | 29.4 | 20.0
  Erythema, Grade 2 (Moderate) | 33.3 | 70.6 | 64.7 | 60.0
  Erythema, Grade 3 (Severe) | 0 | 5.9 | 5.9 | 13.3
  Itching, Grade 0 (None) | 100.0 | 88.2 | 76.5 | 80.0
  Itching, Any Severity >Grade 0 | 0 | 11.8 | 23.5 | 20.0
  Itching, Grade 1 (Mild) | 0 | 11.8 | 23.5 | 20.0
  Pain, Grade 0 (None) | 38.9 | 41.2 | 64.7 | 53.3
  Pain, Any Severity >Grade 0 | 61.1 | 58.8 | 35.3 | 46.7
  Pain, Grade 1 (Mild) | 61.1 | 52.9 | 35.3 | 40.0
  Pain, Grade 2 (Moderate) | 0 | 5.9 | 0 | 6.7

2. Primary Outcome: Percentage of Participants With Unsolicited Adverse Events (AE) by Maximum Severity
Description: An AE is defined as any untoward medical occurrence in a patient or clinical trial participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. AEs are graded from Grade 0=None to Grade 4=Life threatening. AEs are presented as the percentage of participants experiencing an AE, overall and by severity, using the participant's worst reported severity grade.
Time Frame: 28 Days after each dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Number analyzed (Participants) | 18 | 17 | 17 | 15
percentage of participants
  Any Severity | 83.3 | 76.5 | 88.2 | 80.0
  Grade 1 (Mild) | 22.2 | 35.3 | 52.9 | 53.3
  Grade 2 (Moderate) | 44.4 | 23.5 | 17.6 | 20.0
  Grade 3 (Severe) | 11.1 | 17.6 | 5.9 | 6.7
  Grade 4 (Life Threatening) | 5.6 | 0 | 11.8 | 0

3. Primary Outcome: Percentage of Participants With Solicited Systemic AEs as Reported by the Participant Using a Memory Aid 14 Days After Either Vaccine Dose by Maximum Severity
Description: An AE is defined as any untoward medical occurrence in a patient or clinical trial participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Systemic AEs solicited from the participant using a memory aid included: body temperature, headache, myalgia (muscle pain), arthralgia (joint pain), photophobia (sensitivity to light), fatigue (tiredness), body rash, nausea and vomiting. Systemic AEs were graded using the scale: Grade 0= none to Grade 4=Life threatening. Systemic reactions are presented as percentage of participants experiencing a reaction, by reaction type, overall and by severity, using the participant's worst reported severity grade. Only categories for which there was at least 1 participant are reported.
Time Frame: 14 days after each dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Number analyzed (Participants) | 18 | 17 | 17 | 15
percentage of participants
  Temperature, Grade 0 (None) | 94.4 | 100.0 | 88.2 | 100.0
  Temperature, Any Severity >Grade 0 | 5.6 | 0 | 11.8 | 0
  Temperature, Grade 1 (Mild) | 5.6 | 0 | 5.9 | 0
  Temperature, Grade 2 (Moderate) | 0 | 0 | 5.9 | 0
  Headache, Grade 0 (None) | 61.1 | 29.4 | 41.2 | 46.7
  Headache, Any Severity >Grade 0 | 38.9 | 70.6 | 58.8 | 53.3
  Headache, Grade 1 (Mild) | 22.2 | 58.8 | 58.8 | 46.7
  Headache, Grade 2 (Moderate) | 16.7 | 11.8 | 0 | 6.7
  Muscle Pain, Grade 0 (None) | 88.9 | 82.4 | 76.5 | 60.0
  Muscle Pain, Any Severity >Grade 0 | 11.1 | 17.6 | 23.5 | 40.0
  Muscle Pain, Grade 1 (Mild) | 5.6 | 17.6 | 23.5 | 40.0
  Muscle Pain, Grade 2 (Moderate) | 5.6 | 0 | 0 | 0
  Joint Pain, Grade 0 (None) | 88.9 | 88.2 | 88.2 | 86.7
  Joint Pain, Any Severity >Grade 0 | 11.1 | 11.8 | 11.8 | 13.3
  Joint Pain, Grade 1 (Mild) | 5.6 | 11.8 | 5.9 | 13.3
  Joint Pain, Grade 2 (Moderate) | 5.6 | 0 | 5.9 | 0
  Eye Pain, Grade 0 (None) | 88.9 | 94.1 | 88.2 | 93.3
  Eye Pain, Any Severity >Grade 0 | 11.1 | 5.9 | 11.8 | 6.7
  Eye Pain, Grade 1 (Mild) | 11.1 | 5.9 | 11.8 | 6.7
  Increased Sensitivity to Light, Grade 0 | 88.9 | 88.2 | 88.2 | 86.7
  Increased Sensitivity to Light, Severity >Grade 0 | 11.1 | 11.8 | 11.8 | 13.3
  Increased Sensitivity to Light, Grade 1 (Mild) | 11.1 | 5.9 | 11.8 | 13.3
  Increased Sensitivity to Light, Grade 2 (Moderate) | 0 | 5.9 | 0 | 0
  Tiredness, Grade 0 (None) | 66.7 | 70.6 | 47.1 | 60.0
  Tiredness, Any Severity >Grade 0 | 33.3 | 29.4 | 52.9 | 40.0
  Tiredness, Grade 1 (Mild) | 16.7 | 23.5 | 41.2 | 40.0
  Tiredness, Grade 2 (Moderate) | 16.7 | 5.9 | 11.8 | 0
  Rash Anywhere on Body, Grade 0 (None) | 94.4 | 88.2 | 82.4 | 93.3
  Rash Anywhere on Body, Any Severity >Grade 0 | 5.6 | 11.8 | 17.6 | 6.7
  Rash Anywhere on Body, Grade 1 (Mild) | 5.6 | 11.8 | 11.8 | 6.7
  Rash Anywhere on Body, Grade 2 (Moderate) | 0 | 0 | 5.9 | 0
  Nausea, Grade 0 (None) | 83.3 | 88.2 | 88.2 | 93.3
  Nausea, Any Severity >Grade 0 | 16.7 | 11.8 | 11.8 | 6.7
  Nausea, Grade 1 (Mild) | 16.7 | 11.8 | 11.8 | 6.7
  Vomiting, Grade 0 (None) | 94.4 | 100.0 | 94.1 | 100
  Vomiting, Any Severity >Grade 0 | 5.6 | 0 | 5.9 | 0
  Vomiting, Grade 1 (Mild) | 5.6 | 0 | 5.9 | 0

4. Primary Outcome: Percentage of Participants With Solicited Local AEs as Reported by the Participant Using a Memory Aid 14 Days After Either Vaccine Dose by Maximum Severity
Description: An AE is defined as any untoward medical occurrence in a patient or clinical trial participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Local injection site AEs solicited from the participant using a memory aid included: erythema (redness), edema/induration (swelling), pain and pruritus (itching). Local injection site reactions are presented as the percentage of participants experiencing a reaction, by reaction type, overall and by severity, using the participant's worst reported severity grade.
Time Frame: 14 days after each dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Number analyzed (Participants) | 18 | 17 | 17 | 15
percentage of participants
  Swelling, Grade 0 (None) | 50.0 | 41.2 | 35.3 | 40.0
  Swelling, Any Severity >Grade 0 | 50.0 | 58.8 | 64.7 | 60.0
  Swelling, Grade 1 (Mild) | 44.4 | 47.1 | 47.1 | 40.0
  Swelling, Grade 2 (Moderate) | 5.6 | 11.8 | 17.6 | 20.0
  Redness, Grade 0 | 22.2 | 0 | 0 | 20.0
  Redness, Any Severity >Grade 0 | 77.8 | 100 | 100.0 | 80.0
  Redness, Grade 1 (Mild) | 44.4 | 29.4 | 23.5 | 13.3
  Redness, Grade 2 (Moderate) | 33.3 | 64.7 | 64.7 | 46.7
  Redness, Grade 3 (Severe) | 0 | 5.9 | 11.8 | 20.0
  Itching, Grade 0 (None) | 66.7 | 82.4 | 47.1 | 73.3
  Itching, Any Severity >Grade 0 | 33.3 | 17.6 | 52.9 | 26.7
  Itching, Grade 1 (Mild) | 33.3 | 11.8 | 52.9 | 26.7
  Itching, Grade 2 (Moderate) | 0 | 5.9 | 0 | 0
  Pain, Grade 0 (None) | 72.2 | 52.9 | 76.5 | 33.3
  Pain, Any Severity >Grade 0 | 27.8 | 47.1 | 23.5 | 66.7
  Pain, Grade 1 (Mild) | 27.8 | 47.1 | 23.5 | 66.7

5. Primary Outcome: Percentage of Participants With Unsolicited Vaccine-Related AEs Within 28 Days After Either Vaccine Dose by Maximum Severity
Description: An AE is defined as any untoward medical occurrence in a patient or clinical trial participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. AEs are graded from Grade 0=None to Grade 4=Life threatening. AEs are presented as the percentage of participants experiencing an AE causally related to the study treatment as assessed by the investigator, overall and by severity, using the participant's worst reported severity grade. Only categories for which there was at least 1 participant are reported.
Time Frame: 28 Days after each dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Number analyzed (Participants) | 18 | 17 | 17 | 15
percentage of participants
  Any Severity | 16.7 | 17.6 | 52.9 | 33.3
  Grade 1 (Mild) | 11.1 | 11.8 | 41.2 | 33.3
  Grade 2 (Moderate) | 5.6 | 0 | 11.8 | 0
  Grade 3 (Severe) | 0 | 5.9 | 0 | 0

6. Primary Outcome: Percentage of Participants With Abnormal Laboratory Values Reported as Adverse Events (AEs)
Description: The percentage of participants with any clinically relevant abnormal safety laboratory values (chemistry, hematology and urinalysis) collected from vaccine dose 1 (Day 0) through 28 days after dose 2 (Day 90) that were reported as AEs.
  Abnormal laboratory values were reported as AEs based on the following criteria: Grade 3 (Severe) or Grade 4 (Life threatening) laboratory abnormalities based on DMID toxicity tables or laboratory abnormalities which resulted in a medical intervention.
Time Frame: 118 Days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Number analyzed (Participants) | 18 | 17 | 17 | 15
percentage of participants
  Alanine aminotransferase increased | 5.6 | 0 | 0 | 0
  Aspartate aminotransferase increased | 5.6 | 0 | 5.9 | 0
  Blood bilirubin increased | 5.6 | 0 | 0 | 0
  Blood creatine phosphokinase increased | 5.6 | 11.8 | 11.8 | 0
  Occult blood | 0 | 0 | 5.9 | 0

7. Primary Outcome: Seroconversion Rates (SCR) for Each of the Four Dengue Serotypes After First Injection
Description: Seroconversion rate is defined as the percentage of participants with PRNT50 titer ≥ 10 or, if the titer on Day 0 is greater than 10, a four-fold rise in antibody titer.
Time Frame: Day 28
Population: Per Protocol Set included all randomized participants who completed the study without any major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Number analyzed (Participants) | 16 | 13 | 16 | 13
percentage of participants
  DEN-1 | 75.0 [47.6 to 92.7] | 38.5 [13.9 to 68.4] | 62.5 [35.4 to 84.8] | 84.6 [54.6 to 98.1]
  DEN-2 | 62.5 [35.4 to 84.8] | 61.5 [31.6 to 86.1] | 50.0 [24.7 to 75.3] | 76.9 [46.2 to 95.0]
  DEN-3 | 56.3 [29.9 to 80.2] | 23.1 [5.0 to 53.8] | 31.3 [11.0 to 58.7] | 46.2 [19.2 to 74.9]
  DEN-4 | 31.3 [11.0 to 58.7] | 23.1 [5.0 to 53.8] | 50.0 [24.7 to 75.3] | 38.5 [13.9 to 68.4]

8. Primary Outcome: Seroconversion Rates (SCR) for Each of the Four Dengue Serotypes After Second Injection
Description: as for outcome 7
Time Frame: Day 118
Population: Per Protocol Set included all randomized participants who completed the study without any major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Number analyzed (Participants) | 16 | 13 | 16 | 13
percentage of participants
  DEN-1 | 75.0 [47.6 to 92.7] | 69.2 [38.6 to 90.9] | 87.5 [61.7 to 98.4] | 84.6 [54.6 to 98.1]
  DEN-2 | 68.8 [41.3 to 89.0] | 69.2 [38.6 to 90.9] | 62.5 [35.4 to 84.8] | 84.6 [54.6 to 98.1]
  DEN-3 | 75.0 [47.6 to 92.7] | 69.2 [38.6 to 90.9] | 87.5 [61.7 to 98.4] | 84.6 [54.6 to 98.1]
  DEN-4 | 31.3 [11.0 to 58.7] | 30.8 [9.1 to 61.4] | 81.3 [54.4 to 96.0] | 53.8 [25.1 to 80.8]

9. Secondary Outcome: Geometric Mean Titers of Neutralizing Antibody Titers Against Each of the Four Dengue Serotypes
Time Frame: Days 0, 28, 90, 118 and 270
Population: Per Protocol Set included all randomized participants who completed the study without any major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Number analyzed (Participants) | 16 | 13 | 16 | 13
titer
  Day 0 DEN-1 | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  Day 0 DEN-2 | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  Day 0 DEN-3 | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  Day 0 DEN-4 | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  Day 28 DEN-1 | 28.3 [13.0 to 61.3] | 10.5 [4.5 to 24.9] | 27.1 [12.5 to 58.7] | 29.0 [12.3 to 68.6]
  Day 28 DEN-2 | 293.4 [48.0 to 1792.9] | 311.6 [41.8 to 2320.7] | 146.7 [24.0 to 896.5] | 1006.9 [135.2 to 7499.7]
  Day 28 DEN-3 | 32.2 [13.2 to 78.7] | 11.1 [4.1 to 30.0] | 10.0 [4.1 to 24.4] | 19.0 [7.0 to 51.1]
  Day 28 DEN-4 | 13.5 [5.0 to 36.4] | 11.7 [3.9 to 35.2] | 32.2 [12.0 to 86.7] | 20.0 [6.7 to 60.0]
  Day 90 DEN-1 | 29.5 [11.8 to 73.9] | 26.1 [9.4 to 72.2] | 28.9 [11.6 to 72.3] | 19.0 [6.9 to 52.4]
  Day 90 DEN-2 | 174.5 [41.3 to 736.7] | 311.6 [63.0 to 1540.0] | 60.4 [14.3 to 254.9] | 560.1 [113.3 to 2768.5]
  Day 90 DEN-3 | 30.2 [13.5 to 67.3] | 22.3 [9.1 to 54.2] | 11.9 [5.3 to 26.5] | 19.0 [7.8 to 46.2]
  Day 90 DEN-4 | 7.1 [3.4 to 14.8] | 11.7 [5.2 to 26.6] | 20.9 [10.0 to 43.7] | 19.0 [8.4 to 43.0]
  Day 118 DEN-1 | 25.9 [11.8 to 56.9] | 21.1 [8.8 to 50.4] | 60.4 [27.5 to 132.3] | 21.1 [8.8 to 50.4]
  Day 118 DEN-2 | 160.0 [40.1 to 638.3] | 220.3 [47.5 to 1022.7] | 89.2 [22.3 to 355.7] | 429.1 [92.4 to 1991.5]
  Day 118 DEN-3 | 30.8 [15.9 to 60.0] | 19.0 [9.1 to 39.7] | 36.7 [18.9 to 71.3] | 32.3 [15.5 to 67.6]
  Day 118 DEN-4 | 8.4 [4.0 to 17.7] | 10.8 [4.7 to 24.8] | 54.2 [25.7 to 114.3] | 22.3 [9.7 to 51.0]
  Day 270 DEN-1 | 16.8 [8.2 to 34.6] | 12.4 [5.6 to 27.5] | 24.8 [12.1 to 51.1] | 10.5 [4.7 to 23.5]
  Day 270 DEN-2 | 118.1 [32.2 to 433.0] | 173.3 [41.0 to 732.2] | 54.2 [14.8 to 198.5] | 265.5 [62.9 to 1121.8]
  Day 270 DEN-3 | 21.8 [12.0 to 39.5] | 14.5 [7.5 to 28.1] | 14.8 [8.2 to 26.7] | 14.5 [7.5 to 28.1]
  Day 270 DEN-4 | 8.4 [4.5 to 15.8] | 10.0 [5.0 to 20.1] | 28.3 [15.1 to 53.1] | 13.8 [6.9 to 27.7]

10. Secondary Outcome: Seroconversion Rates (SCR) for Each of the Four Dengue Serotypes at Days 90 and 270
Description: as for outcome 7
Time Frame: Days 90 and 270
Population: Per Protocol Set included all randomized participants who completed the study without any major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Number analyzed (Participants) | 16 | 13 | 16 | 13
percentage of participants
  Day 90 DEN-1 | 68.8 [41.3 to 89.0] | 61.5 [31.6 to 86.1] | 62.5 [35.4 to 84.8] | 76.9 [46.2 to 95.0]
  Day 90 DEN-2 | 75.0 [47.6 to 92.7] | 69.2 [38.6 to 90.9] | 43.8 [19.8 to 70.1] | 84.6 [54.6 to 98.1]
  Day 90 DEN-3 | 62.5 [35.4 to 84.8] | 61.5 [31.6 to 86.1] | 43.8 [19.8 to 70.1] | 61.5 [31.6 to 86.1]
  Day 90 DEN-4 | 18.8 [4.0 to 45.6] | 30.8 [9.1 to 61.4] | 56.3 [29.9 to 80.2] | 46.2 [19.2 to 74.9]
  Day 270 DEN-1 | 62.5 [35.4 to 84.8] | 46.2 [19.2 to 74.9] | 75.0 [47.6 to 92.7] | 61.5 [31.6 to 86.1]
  Day 270 DEN-2 | 62.5 [35.4 to 84.8] | 69.2 [38.6 to 90.9] | 50.0 [24.7 to 75.3] | 84.6 [54.6 to 98.1]
  Day 270 DEN-3 | 68.8 [41.3 to 89.0] | 53.8 [25.1 to 80.8] | 75.0 [47.6 to 92.7] | 69.2 [38.6 to 90.9]
  Day 270 DEN-4 | 25.0 [7.3 to 52.4] | 23.1 [5.0 to 53.8] | 75.0 [47.6 to 92.7] | 46.2 [19.2 to 74.9]

11. Secondary Outcome: Percentage of Participants With Serotype-Specific DENVax RNA Detected Due to Each of the Four Dengue Vaccine Components After Each Vaccination
Description: A quantitative reverse transcriptase-polymerase chain reaction (qRT-PCR) assay was used for detection and serotype identification of dengue viral ribonucleic acid (RNA) that is present in serum. A test for viremia is considered positive if the assay value is >= 3.6, which is the limit of quantification (LOQ), negative if the assay value was zero, and undetermined if the assay value is >0 but <3.6. The percentage of participants with positive results is reported.
Time Frame: Day 0 to Day 104
Population: Full analysis set included all randomized participants who received at least one dose of study vaccine and for whom valid pre-dosing and at least one valid sample for immunogenicity (eg, seroconversion) was received.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Number analyzed (Participants) | 18 | 17 | 17 | 15
percentage of participants
  DEN-1 | 0 | 0 | 0 | 0
  DEN-2 | 38.9 | 23.5 | 23.5 | 53.3
  DEN-3 | 5.6 | 5.9 | 0 | 0
  DEN-4 | 0 | 0 | 0 | 0

12. Primary Outcome: Percentage of Participants With Unsolicited Vaccine-Related SAEs
Description: A serious adverse event (SAE) is any AE in the view of the investigator that results in any of the following outcomes: death, life threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that may require medical or surgical intervention to prevent one of the other serious outcomes.
Time Frame: Dose 1 until 28 days after Dose 2 (Up to Day 118)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Number analyzed (Participants) | 18 | 17 | 17 | 15
percentage of participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited Adverse Events: 28 days after either vaccination. Serious Adverse Events: Dose 1 until 28 days after Dose 2 (Up to Day 118).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Events meeting the protocol-specified seriousness criteria were reported as SAEs.
Arm/Group | Group 1: TDV Using PharmaJet® Injector | Group 2: TDV Using PharmaJet® Injector | Group 3: TDV Using Needle and Syringe | Group 4: TDV Using PharmaJet® Injector
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 15/18 | 13/17 | 15/17 | 12/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: TDV Using PharmaJet® Injector (N=18) | Group 2: TDV Using PharmaJet® Injector (N=17) | Group 3: TDV Using Needle and Syringe (N=17) | Group 4: TDV Using PharmaJet® Injector (N=15)
Injection site haematoma (General disorders) | 2 | 0 | 3 | 0
Injection site warmth (General disorders) | 0 | 0 | 0 | 3
Vessel puncture site haematoma (General disorders) | 2 | 1 | 1 | 0
Vessel puncture site pain (General disorders) | 1 | 1 | 2 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 4 | 3
Urinary tract infection (Infections and infestations) | 3 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 2 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0
Injection site discolouration (General disorders) | 0 | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 1 | 1
Injection site pain (General disorders) | 1 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Chlamydial infection (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Gingival infection (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 2
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Occult blood (Investigations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days. The sponsor is permitted to protect any proprietary information and to provide comments based on information from other studies that may not be available to the Investigator.